CLINICAL TRIAL: NCT00002244
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Pivotal Clinical Study Evaluating the Safety and Efficacy of WF10 (TCDO) Intravenous Solution in the Management of Patients With Late-Stage HIV Disease
Brief Title: A Study to Evaluate the Safety and Effectiveness of WF10 Given to Patients With Late-Stage HIV Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OXO Chemie (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 222C
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: HIV Infections
Keywords: Placebos; Infusions, Intravenous; Quality of Life; Anti-HIV Agents; tetrachlorodecaoxide
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: WF10

SUMMARY:
The purpose of this study is to see if it is safe and effective to give WF10 to adults with late-stage HIV disease. WF10 is suspected to help the immune system fight infection and slow HIV disease progression.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 treatment groups to receive 4 IV treatment cycles of either WF10 or control (physiological saline solution). Patients are monitored throughout the study for: a) clinical progression; b) number, duration, and cause of hospitalizations; c) quality of life; and d) density of CD38 antigen on CD8+ T cells. Patients receive treatment for 11 weeks but will continue to be followed for a maximum of 96 weeks. During the follow-up period, patients are evaluated initially at Week 18, then at Weeks 24, 36, and 48. If the study is continued beyond Week 48, follow-up visits are conducted at Weeks 72 and 96.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a CD4 cell count of less than 50 cells/mm3 within 14 days prior to study entry.
* Are at least 18 years old.
* Have received anti-HIV drugs at some time in the past.
* Agree to practice abstinence or use effective methods of birth control, including the pill, during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are being treated for any form of cancer within 30 days of study entry.
* Have ever received an HIV vaccine.
* Have received steroids within 30 days prior to study entry. (Note: Testosterone is allowed.)
* Have received certain medications, including anti-HIV treatments that are not approved by the FDA.
* Have participated in another WF10 study.
* Have an illness or any condition that might exclude them from this study.
* Are pregnant or breast-feeding.
* Abuse drugs or medications.
* Received a blood transfusion within 45 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240

CONTACTS AND LOCATIONS:
Locations (32):
- United States (27):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Tower Infectious Disease Med Ctr, Los Angeles, California
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - ViRx Inc, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - Ctr for Quality Care, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Leahi Hosp / Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Med Ctr / Section of Infectious Diseases, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Univ of Iowa Hosp & Clinic, Iowa City, Iowa
  - Boston Med Ctr / Clinical Research Office, Boston, Massachusetts
  - Univ Health Ctr, Detroit, Michigan
  - Regions Hosp, Saint Paul, Minnesota
  - Truman Med Ctr / Infectious Disease Clinic, Kansas City, Missouri
  - Newark Community Health Ctr, Newark, New Jersey
  - Univ of New Mexico Health Science Center, Albuquerque, New Mexico
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - MCP Hahnemann Univ, Philadelphia, Pennsylvania
  - Ludwig Lettau Private Practice, Charleston, South Carolina
  - Burnside Clinic, Columbia, South Carolina
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Virginia Mason Research Center / Clinical Trial Unit, Seattle, Washington
- Canada (5):
  - St Paul's Hosp, Vancouver, British Columbia
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Ottawa General Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Montreal Gen Hosp / Div of Clin Immuno and Allergy, Montreal, Quebec